CLINICAL TRIAL: NCT06016049
Title: Cerebral Changes Following Carpal Tunnel Syndrome Treated With Guided Brain Plasticity
Brief Title: Cerebral Changes Following CTS Treated With Guided Plasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 210817
Record Dates: First submitted 2023-06-11; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Magnetic Resonance Imaging; Somatosensory Cortex; Anesthesia; Hand
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- EMLA® (Active Comparator): adjuvant forearm anesthesia cream (EMLA®) and sensibility training in a program involving 15 sessions (8 weeks) of guided plasticity
  Interventions: Other: EMLA® adjuvant; Behavioral: Sensory training
- Skin cream (Placebo Comparator): skin cream and sensibility training in a program involving 15 sessions (8 weeks) of guided plasticity training
  Interventions: Behavioral: Sensory training

INTERVENTIONS:
Other: EMLA® adjuvant — cutaneous forearm deafferentation
  Arms: EMLA®
Behavioral: Sensory training — Sensibility training of the median nerve

SUMMARY:
70 patients with mild to moderate Carpal tunnel Syndrome (CTS) including 24 patients with unilateral CTS were randomized to treatment with ipsilateral cutaneous forearm deafferentation with an anesthetic cream (EMLA®) or placebo during 8 weeks. Patient-rated outcomes was assessed using the symptom severity scale from the Boston carpal tunnel syndrome questionnaire (BCTQ) and the disability of arm, shoulder and hand questionnaire(Quick-DASH). Clinically patients were assessed for tactile discrimination and dexterity and nerve conduction studies (NCS). Cortical activation during sensory stimulation was evaluated with functional magnetic resonance imaging (fMRI) at 3T. Assessments were performed at baseline, after 90 min of initial treatment, and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of CTS for more than 3 months
* classic or probable CTS according to Katz' hand diagram (2, 27)
* clinical signs of unilateral CTS with a positive Tinel's and Phalen's test
* age between 18 and 70 years
* nerve conduction studies (NCS) with a fractionated sensory nerve conduction velocity for the median nerve across the wrist of 40 m/s or less on the affected side and of more than 43 m/s on the contralateral side
* no contraindications for MR examinations.

Exclusion Criteria:

* bilateral symptoms
* having been operated for CTS previously
* prior wrist or carpal fracture
* diabetes
* thyroid disease
* rheumatoid arthritis
* neurological disease
* drug abuse
* complete conduction block on electroneurography or prior regular exposure to hand-held vibrating tools.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Symptom Severity Score | 8 weeks
  score between 1 and 5, with higher scores indicating worse symptoms or function
functional MRI activation affected vs healthy side (more activation voxels means more active brain area) | 8 weeks
  The difference in activation using interaction contrast between baseline vs 8 weeks in somatosensory cortex (affected vs healthy side)

SECONDARY OUTCOMES:
quick-DASH upper extremity symptom score | 8 weeks
  score between 1-5, higher scores indicating less symptoms
2 Point Discrimination (2PD) | 8 weeks
  mean value of 3 measures indicating touch threshold
Sensory conduction velocity | 8 weeks
  Sensory Nerve Conduction Velocity from nerve conduction studies
Sensory conduction amplitude | 8 weeks
  Sensory Nerve Conduction Amplitude from nerve conduction studies
functional MRI dig 1+2 | 8 weeks
  comparison between activation using interaction contrast in S1sensory cortex of the
functional MRI dig 5 | 8 weeks
  comparison between activation in the sensory cortex of the little finger (EMLA® vs placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Flondell, MD PhD, Principal Investigator — Institute of Translational Sciences Malmö, Lund University; Anders Björkman, MD, Prof., Study Chair — Institute of Clinical Sciences, Sahlgrenska Academy, Gothenburg University

IPD SHARING:
Plan to Share IPD: No
data can be shared upon reasonable demand after personal contact.